CLINICAL TRIAL: NCT02380651
Title: Functional Outcomes and Health Related Quality of Life in Upper-extremity Sarcoma Patients After Limb Salvage: a Prospective Study
Brief Title: Functional Outcomes and HRQoL in Upper-extremity Sarcoma Patients After Limb Salvage
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Jussi Repo, MD, Helsinki University Central Hospital
Other Study IDs: 324/13/03/02/2014/1
Record Dates: First submitted 2015-03-01; First posted 2015-03-05 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Cancer of Muscle
MeSH Terms: conditions — Muscle Neoplasms | interventions — Limb Salvage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Limb salvage — Local or free flaps

SUMMARY:
This study aims to assess the functional ability and health-related quality of life (HRQoL) of upper extremity sarcoma patients who have undergone limb salvage surgery.

DETAILED DESCRIPTION:
The purpose of this study is to assess the functional capabilities and health-related quality of life (HRQoL) of upper-extremity sarcoma patients who have undergone limb salvage surgery.

Patient hospital records are retrospectively reviewed for demographic and clinical data.

The patient recruitment takes place at the outpatient clinic of the Comprehensive Cancer Center, Helsinki University Hospital, and Tampere University Hospital. The study includes a cross-sectional assessment at six months follow-up with five validated questionnaires. A follow-up is conducted two and five years after surgery in the outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Upper extremity soft tissue sarcoma locating in between scapula to arm
* No metastasis at the time of diagnosis
* Undergone limb salvage surgery
* A minimum of 6 months follow-up
* Written consent
* Age > 18

Exclusion Criteria:

* Age <18
* No limb-salvage surgery due to sarcoma
* Deceased

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Upper extremity sarcoma patient who underwent limb-salvage surgery
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-12; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life and upper-extremity functional capability | 6 months to five years
  To assess health-related quality of life and upper-extremity functional capability

SECONDARY OUTCOMES:
Sarcoma recurrence | 6 months to five years
  to assess sarcoma recurrence
Quality of Life Questionnaire-Core 30 | 6 months to five years
  to assess the health-related quality of life
the 15D health-related quality of life instrument | 6 months to five years
  to assess the health-related quality of life
The QuickDASH | 6 months to five years
  to assess the upper-extremity function
The MSTS upper extremity section | 6 months to five years
  to assess the upper-extremity function
The TESS upper extremity section | 6 months to five years
  to assess the upper-extremity function

OTHER OUTCOMES:
Visual Analogue Scale for pain | 6 months to five years
  to assess pain

CONTACTS AND LOCATIONS:
Overall Officials: Erkki J Tukiainen, MD, PhD, Study Director — Helsinki University Central Hospital; Carl Blomqvist, MD, PhD, Study Director — Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Helsinki University Central Hospital, Helsinki, Uusimaa
  - Tampere University Hospital, Tampere